CLINICAL TRIAL: NCT00451607
Title: Evaluation of Environmental Stress and Individualized Sensorimotor Care on Autonomic Nervous System Activity in a Premature Population : a Prospective Study
Brief Title: Environmental Stress and Individualized Sensorimotor Care on Autonomic Nervous System Activity in Premature Population
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint Etienne
Other Study IDs: SNA STRESS 07
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Premature Birth
Keywords: premature; newborn; heart rate variability; individualized sensorimotor care; noise
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Autonomic nervous system (ANS) is an essential regulator for the homeostasis, circulatory and respiratory systems. Heart rate variability, under the dependence of the parasympathetic and orthosympathetic arms is a peripheral witness of its well functioning.

Activity ANS indices are technically measurable from the birth by non invasive cardiac monitoring: in given environmental conditions. According to the individualized care given to the baby, we can easily observe by frequential analysis, modifications of ANS level activity; If for a full-term newborn, the balance of ANS allows him to adapt its cardiac frequency to its internal and external environment (thermoregulation, baroreflex, sinus arrhythmia, awakening state) , the premature birth is at the origin of a prolonged defect of global ANS maturation, probably induced by external environmental and stress factors (pain, stimulations, aggressive noise and lights). This disrupted maturation profile in case of prematurity, was confirmed in two preliminary studies on premature babies reaching term for gestational age.

We hypothesis that adapted sensorimotor care could decrease this stress and optimize the ANS activity profile.

In a prospective study, by a non invasive real-time measure, we analyse impact of stress on ANS activity in a premature population, hospitalized in our neonatal intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* premature birth
* hospitalized in the intensive care unit or in the neonatology unit or in the reanimation unit of the Pediatric Hospital of SAINT-ETIENNE

Exclusion Criteria:

* arrhythmias
* general anaesthesia three weeks before the records

Ages: 1 Day to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature Birth
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Patural H, Barthelemy JC, Pichot V, Mazzocchi C, Teyssier G, Damon G, Roche F. Birth prematurity determines prolonged autonomic nervous system immaturity. Clin Auton Res. 2004 Dec;14(6):391-5. doi: 10.1007/s10286-004-0216-9. PMID 15666067
- [Result] Patural H, Pichot V, Jaziri F, Teyssier G, Gaspoz JM, Roche F, Barthelemy JC. Autonomic cardiac control of very preterm newborns: a prolonged dysfunction. Early Hum Dev. 2008 Oct;84(10):681-7. doi: 10.1016/j.earlhumdev.2008.04.010. Epub 2008 Jun 16. PMID 18556151